CLINICAL TRIAL: NCT04809402
Title: Cataract Online Refraction Evaluation: A Multi Center Randomized Controlled Trial
Acronym: CORE-RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: Health Holland (Other)
Responsible Party: Principal Investigator, Robert P.L. Wisse, MD PhD, Principal Investigator, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NL74625.041.20
Record Dates: First submitted 2021-03-10; First posted 2021-03-22 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Cataract
Keywords: e-health; digital; remote monitoring
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemonitoring (Other): Subjects in the telemonitoring group will have post-operative follow-up measurements involving teleconsultations, remote eye exams and health questionnaires.
  Interventions: Other: remote monitoring after cataract surgery
- Usual care (No Intervention): Subjects in the usual care group will receive regular post-operative care, mostly involving in-hospital consultations.

INTERVENTIONS:
Other: remote monitoring after cataract surgery — remote monitoring after cataract surgery
  Arms: Telemonitoring

SUMMARY:
Background of the study:

Cataract is widely prevalent in especially elderly and cataract extraction surgery has thus become one of the most performedsurgeries worldwide. In recent decades the safety of cataract surgery has greatly improved and it is considered one of the safestsurgeries to be performed. Postoperative management consists of routine examinations within one week, to ascertain no adverseevents have occurred immediately after surgery, and between 4-6 weeks, to determine the refractive error. The incidence of seriousadverse events following cataract surgery is estimated to be 1%. As a result, the majority of patient visits after cataract surgery willbe uneventful. Nonetheless valuable time and hospital resources are consumed. Remote monitoring could replace clinicalexaminations in selected patient groups. However, this practice of digital remote monitoring which the patient can use independentlyhas not been clinically validated yet.

Objective of the study:

To determine non-inferiority of the corrected distance visual acuity (CDVA) with the prescription obtained through the web-basedmeasurement of refractive error, compared to usual care, in patients who underwent routine cataract surgery.

Study design:

Observational randomized trial without interventions

Study population:

Patients eligible for cataract surgery, without visual acuity influencing comorbidities or predisposing complicating factors.

Primary study parameters/outcome of the study:

costeffectiveness

Secundary study parameters/outcome of the study (if applicable):

Corrected distance visual acuity at the final post-operative visit, uncorrected distance visual acuity, refractive error(sphere/cylinder/axes), patient reported outcome measurements, adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Planned for bilateral phacoemulsification cataract extraction and intra-ocular lens implantation (either sequentialor in one procedure)
* ≥ 18 years of age
* No other current ophthalmic conditions or history that negatively influence post-operative visual acuity
* Be able to fill out the health questionnaires (in Dutch, German or English) and perform the web-based refractiveassessment (possibly with assistance of family member or other close relative).
* Specific digital requirements include access to a computer and a smartphone and knowledge how to log in to anonline patient portal.

Exclusion Criteria:

* Cataract extraction surgery combined with other procedures, including: keratoplasty, vitrectomy, glaucoma filter implants
* Ocular comorbidities that negatively influence post-operative visual acuity
* No access to the digital requirements to take the online health questionnaire and/or perform the online refraction.
* Insufficient command of the Dutch, German or English language to understand the questionnaires andinstructions of the web-based refractive assessment or no family member / close relative to assist with this
* Inability of performing the web-based eye exam prior to cataract surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-07-22 (Estimated)

PRIMARY OUTCOMES:
Cost-effectiveness | pre-operative until 3 months after surgery
  The main outcome measure will be Incremental cost-effectiveness ratio (ICER), defined as euros per QALY, and compared between the two groups.

SECONDARY OUTCOMES:
Corrected distance visual acuity at the final post-operative visit (achieved with web-based vs manifest refraction) | 4-6 weeks after surgery
  The corrected distance visual acuity achieved with the web-based refraction will be compared to the corrected distance visual acuity that is achieved with the subjective refraction.
Uncorrected distance visual acuity (web-based vs reference chart) | pre-operative, 4-6 weeks after surgery
  The uncorrected distance visual acuity that is assessed in the web-based assessment will be compared to the uncorrected distance visual acuity that is assessed using the reference chart.
Refractive error in sphere/cylinder/axes (web-based vs reference chart) | 4-6 weeks after surgery
  The refractive error (in sphere/cylinder/axes) will be asssessed by the web-based assessment and compared to the subjective refractive error assessment.
Patient reported outcomes | pre-operative vs 3 months after surgery
  The PROMs questionnaire (CatQuest-9SF) assesses the patient's own reported visual disability from cataract and the improvement after surgery. High scores represent better visual acuity. The results of the PROMs questionnaire will be compared between the groups to assess differences and determine if a web-based follow-up strategy influences these subjective measures. PROMs will be offered in Dutch, German or English accordingly and assessed at baseline and at 3 months follow-up.
Adverse events / additional consultations | pre-operative until 3 months after surgery
  All unplanned additional consultations (telephone or hospital) will be recorded. We will count these and compare the frequencies between the two groups.
Total costs | pre-operative until 3 months after surgery
  Total costs (in euros) will be determined for both groups. We will count costs for hospital resources and staff, as well as costs for the patient (such as travel and parking costs).
QALY's | pre-operative and 3 months after surgery
  To determine the QALY, patients of both groups will be requested to fill out questionnaires to assess quality of life (EQ-5D). A unique health state is defined by combining one level from each of the five dimensions. Higher levels indicate more problems.

CONTACTS AND LOCATIONS:
Locations (6):
- Vienna Institute for Research in Ocular Surgery, Austria, Vienna, Austria
- Augenklink Sulzbach, Sulzbach, Germany
- Netherlands (4):
  - Amphia Ziekenhuis, Breda, North Brabant
  - Oogcentrum Noordholland, Heerhugowaard, North Holland
  - Maastricht UMC+, Maastricht
  - Janneau Claessens, Utrecht

REFERENCES:
- [Derived] Claessens JLJ, Wanten JC, Bauer NJC, Nuijts RMMA, Vrijman V, Selek E, Wouters RJ, Reus NJ, van Dorst FJGM, Findl O, Ruiss M, Boden K, Januschowski K, Imhof SM, Wisse RPL. Web-based telemonitoring of visual function and self-reported postoperative outcomes in cataract care: international multicenter randomized controlled trial. J Cataract Refract Surg. 2024 Sep 1;50(9):947-955. doi: 10.1097/j.jcrs.0000000000001492. PMID 38809014
- [Derived] Claessens JLJ, Maats EPE, Iacob ME, Wisse RPL, Jongsma KR. Introducing e-health technology to routine cataract care: patient perspectives on web-based eye test for postoperative telemonitoring. J Cataract Refract Surg. 2023 Jul 1;49(7):659-665. doi: 10.1097/j.jcrs.0000000000001189. Epub 2023 Mar 29. PMID 37010267
- [Derived] Claessens JLJ, Wanten JC, Bauer NJC, Nuijts RMMA, Findl O, Huemer J, Imhof SM, Wisse RPL. Remote follow-up after cataract surgery (CORE-RCT): study protocol of a randomized controlled trial. BMC Ophthalmol. 2023 Jan 30;23(1):41. doi: 10.1186/s12886-023-02779-7. PMID 36717799